CLINICAL TRIAL: NCT00530218
Title: Phase II Study of Intravenous Ganciclovir Followed by Oral Ganciclovir in the Treatment of Reactivation of CMV Following Bone Marrow Transplant
Brief Title: Ganciclovir by Infusion and by Mouth in Treating Patients With Cytomegalovirus After Donor Bone Marrow Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 98074; P30CA033572 (NIH); CHNMC-98074 (Other: City of Hope National Medical Center); CDR0000564546 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Leukemia; Lymphoma; Multiple Myeloma; MDS; Myelodysplastic/Myeloproliferative Diseases
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic-Myeloproliferative Diseases | interventions — Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Study Participants (Experimental): Ganciclovir IV 5 mg/kg/bid x 7 days followed by Ganciclovir Oral 1000 mg tid 7 days per week x 5 weeks
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir — Following the first CMV-positive blood culture on day 21 or later, or the first two consecutive CMV-positive PCR tests on day 21 or later, 5mg/kg/bid x 7 days of Ganciclovir is given intravenously, followed by oral Ganciclovir 1000 mg tid 7 days per week x 5 weeks
  Other Names: Cytovene

SUMMARY:
RATIONALE: Antiviral drugs, such as ganciclovir, act against viruses. Giving ganciclovir by infusion and then by mouth may be effective treatment for cytomegalovirus that has become active after donor bone marrow transplant.

PURPOSE: This phase II trial is studying how well giving ganciclovir by infusion and by mouth works in treating patients with cytomegalovirus after donor bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility of using oral ganciclovir (GCV) following induction with intravenous GCV in the setting of cytomegalovirus (CMV) reactivation after bone marrow transplantation.

OUTLINE: Blood cultures for cytomegalovirus (CMV) are obtained periodically after the planned bone marrow transplantation (BMT). Patients showing reactivation of CMV receive induction ganciclovir (GCV) IV twice a day on days 1-7. Patients then receive maintenance oral GCV three times a day for 5 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Undergoing allogeneic transplantation, including unrelated donor bone marrow transplantation (BMT) and/or allogeneic donor leukocyte infusion, for any indication
* Patients or their donors must have had a positive pre-BMT cytomegalovirus (CMV) antibody titer as measured by enzyme-linked immunosorbent assay (ELISA)

PATIENT CHARACTERISTICS:

* Able to comply with study requirements

Exclusion criteria:

* Signs or symptoms of documented CMV infection, including any positive CMV culture from any site and/or any suspected or documented CMV-associated clinical syndrome, at the time of study entry
* History of symptomatic CMV-associated clinical syndrome

PRIOR CONCURRENT THERAPY:

* Receiving concurrent investigational antiviral agents

PATIENT CHARACTERISTICS:

* History of hypersensitivity to ganciclovir or acyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1999-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo T. Spielberger, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope National Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] R. Spielberger, J. Zaia, R. A. Nelson, E. Newman, G. Gallez-Hawkins, A. Ahlers, J. Stevenson, C. Acedo, A. Alam, R. Bhatia, S. Cohen, P. Falk, H. Fung, A.Kashyap, N. Kogut, Al Krishnan, A. Molina, A. Nademanee, M. O'Donnell, P. Parker, L. Popplewell, R. Rodriguez, F. Sahebi, D. Snyder, A. Stein, S. Forman. Use of Oral Ganciclovir (PO-GCV) for the Preemptive Treatment (Tx) of CMV Following Allogeneic HCT: Safety and Feasibility Results. Blood 96 (11): 586A # 2516, 2000.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Patients undergo intervention with intravenous ganciclovir followed by oral ganciclovir, if cytomegalovirus reactivation is detected.
Period: Overall Study
Arm/Group | All Study Participants
Started | 61
Completed | 36 (CMV Reactivation Was Detected)
Not Completed | 25
Not completed — CMV Not Detected | 13
Not completed — Death | 12

BASELINE CHARACTERISTICS:
Population: All patients start out in the "No CMV Reactivation" period, at least until day 21 when the first blood culture or PCR tests are performed. After one positive blood culture or two consecutive positive PCR tests, patients move to the "CMV Reactivation Detected" period. Tests are performed twice weekly from day 21 post-transplant to day 100.
Groups:
- All Study Participants: Blood Culture at Day 21 or later -or- PCR Test at Day 21 or later
Arm/Group | All Study Participants
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 41 [19 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This will be measured by the number of the CMV+ participants with adverse events occurring when receiving oral GCV.
Time Frame: From first ganciclovir positive test, after day 21 post-hematopoietic cell transplant
Population: Patients are treated with Intravenous Ganciclovir followed by Oral Ganciclovir on detection of CMV reactivation. Among the 36 patients with CMV reactivation, four patients' adverse event data are not available.
Measure: Count of Participants; unit: Participants
Groups:
- CMV Reactivation Patients With GCV: CMV reactivation patients with intravenous Ganciclovir followed by oral Ganciclovir.
Arm/Group | CMV Reactivation Patients With GCV
Number analyzed (Participants) | 32
Participants
  Haptoglobin | 1
  Hemoglobin | 31
  Hemolysis | 1
  Leukocytes | 22
  Lymphopenia | 2
  Neutrophils/granulocytes | 12
  Platelets | 26
  pRBCs | 17
  aGVHD | 21
  cGVHD | 1
  Palpitations | 1
  Supraventricular and nodal arrhythmia | 19
  Cardiac General - Other | 1
  Hypertension | 13
  Hypotension | 5
  Edema | 8
  INR | 1
  Fatigue | 21
  Fever | 10
  Insomnia | 3
  Rigors/Chills | 6
  Sweating | 1
  Weight loss | 3
  Bruising | 2
  Skin - Other | 3
  Dry Skin | 5
  Flushing | 4
  Hair Loss / Alopecia | 4
  Pigmentation Changes | 5
  Pruritus/Itching | 3
  Rash/Desquamation | 3
  Rash/Desquamation w GVHD | 19
  Wound Complication, Non-infection | 1
  Cushingoid Appearance | 15
  Endocrine - Other | 2
  Thyroid Function, Low (Hypothyroidism) | 1
  Anorexia | 15
  Constipation | 1
  Dehydration | 16
  Diarrhea | 4
  Diarrhea with GVHD | 4
  Dry mouth/Salivary Gland (Xerostomia) | 2
  Esophagitis | 2
  Flatulence | 4
  Gastritis | 2
  Gastrointestinal - Other | 6
  Heartburn/Dyspepsia | 4
  Mucositis/Stomatitis | 1
  Nausea | 22
  Stomatitis/pharyngitis (Oral/Pharyngeal Mucositis) | 16
  Taste Alteration (Dysgeusia) | 5
  Vomiting | 14
  Hematuria (in the absence of vaginal bleeding) | 4
  Hemorrhage/bleeding w/ grade 3 or 4 thrombocytopni | 2
  Hemorrhage/bleeding w/o grade 3 or 4 thrombocytope | 2
  Hemorrhage, pulmonary/upper respiratory | 1
  Hemorrhage/Bleeding - Other | 1
  Petechiae/purpura | 1
  Bilirubin with GVHD | 5
  Febrile Neutropenia | 1
  Infection - Other | 1
  Infection w/ unknown ANC | 3
  Infection - Bacterial | 13
  Infection - Fungal | 3
  Infection - Viral | 8
  Lymphatics | 1
  ALT, SGPT | 31
  AST, SGOT | 23
  Albumin, serum-low (hypoalbuminemia) | 25
  Alkaline phosphatase | 11
  Bilirubin (hyperbilirubinemia) | 8
  CPK (creatine phosphokinase) | 1
  Calcium, serum-high (hypercalcemia) | 1
  Calcium, serum-low (hypocalcemia) | 20
  Cholesterol, serum-high (hypercholesteremia) | 23
  Creatinine | 20
  Glucose, serum-high (hyperglycemia) | 24
  Magnesium, serum-high (hypermagnesemia) | 4
  Magnesium, serum-low (hypomagnesemia) | 27
  Metabolic/Laboratory - Other | 1
  Phosphate, serum-low (hypophosphatemia) | 21
  Potassium, serum-high (hyperkalemia) | 7
  Potassium, serum-low (hypokalemia) | 16
  Proteinuria | 1
  Sodium, serum-low (hyponatremia) | 15
  Uric acid, serum-high (hyperuricemia) | 5
  Muscle weakness, generalized or specific area | 3
  Musculoskeletal/Soft Tissue - Other | 2
  Myositis (inflammation/damage of muscle) | 1
  Confusion | 1
  Dizziness | 5
  Memory Impairment | 1
  Mood Alteration | 11
  Neurology - Other | 4
  Neuropathy: Motor | 1
  Neuropathy: Sensory | 3
  Speech Impairment | 1
  Syncope | 1
  Tremor | 12
  Dry eye syndrome | 2
  Ocular/Visual - Other | 4
  Ophthalmoplegia/diplopia (double vision) | 1
  Pain | 25
  Adult Respiratory Distress Syndrome (ARDS) | 2
  Cough | 7
  Dyspnea (shortness of breath) | 7
  Hypoxia | 2
  Pleural effusion (non-malignant) | 1
  Pneumonitis/pulmonary infiltrates | 6
  Pulmonary/Upper Respiratory - Other | 2
  Urinary frequency/urgency | 1
  Urinary retention (including neurogenic bladder) | 1
  Thrombosis/thrombus/embolism | 1

2. Primary Outcome: Observation of Cytomegalovirus (CMV) in Blood as Measured by Either Blood Culture or Polymerase Chain Reaction (PCR) During the Course of Antiviral Treatment
Time Frame: Twice Weekly after day 21 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 61
Participants
  CMV Reactivation | 36
  No CMV Reactivation | 25

3. Primary Outcome: Compliance Rate Among Patients With CMV Reactivation
Description: CMV reactivation patients completed 6-week GCV therapy.
Time Frame: From first ganciclovir positive test to the end of the 6th week GCV therapy
Population: Among the 36 patients with CMV reactivation, two patients are in-evaluable for compliance.
Measure: Number; unit: participants
Groups:
- Compliance Among Patients With CMV Reactivation: Patients with CMV reactivation detected by blood culture or PCR test.
Arm/Group | Compliance Among Patients With CMV Reactivation
Number analyzed (Participants) | 34
participants
  Compliance | 26
  No Compliance | 8

ADVERSE EVENTS:
Time Frame: Death was monitored from Day 0 up to Year 11. Serious and other adverse events were assessed from Day 21 up to Day 100.
Description: Death was monitored for all participants. Adverse events were assessed for the CMV+ participants, who were treated with intravenous Ganciclovir followed by oral Ganciclovir on detection of CMV reactivation. Among the 36 patients with CMV reactivation, four patients' adverse event data are not available.
Groups:
- Patients With CMV Reactivation Detected: CMV Positive Blood Culture at Day 21 or later -or- CMV Positive PCR Test at Day 21 or later
- Patients Without CMV Reactivation Detected: No CMV Positive Blood Culture at Day 21 or later -and- No CMV Positive PCR Test at Day 21 or later
Arm/Group | Patients With CMV Reactivation Detected | Patients Without CMV Reactivation Detected
All-Cause Mortality (participants affected / at risk) | 19/36 | 14/25
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/0
Other Adverse Events (participants affected / at risk) | 32/32 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With CMV Reactivation Detected (N=32) | Patients Without CMV Reactivation Detected (N=0)
Haptoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 31 (31) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 22 (22) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 12 (12) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 26 (26) | 0 (0)
pRBCs (Blood and lymphatic system disorders) | 17 (17) | 0 (0)
Acute graft versus host disease (Blood and lymphatic system disorders) | 21 (21) | 0 (0)
Chronic graft versus host disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 19 (19) | 0 (0)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 13 (13) | 0 (0)
Hypotension (Cardiac disorders) | 5 (5) | 0 (0)
Edema (Cardiac disorders) | 8 (8) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21 (21) | 0 (0)
Fever (General disorders) | 10 (10) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0)
Rigors/chills (General disorders) | 6 (6) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 3 (3) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pigmentation changes (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash/desquamation with GVHD (Skin and subcutaneous tissue disorders) | 19 (19) | 0 (0)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cushingoid appearance (Endocrine disorders) | 15 (15) | 0 (0)
Endocrine - Other (Endocrine disorders) | 2 (2) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 15 (15) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 16 (16) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhea with GVHD (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 6 (6) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (22) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 16 (16) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (14) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Investigations) | 4 (4) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Investigations) | 2 (2) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Investigations) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Investigations) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Investigations) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Investigations) | 1 (1) | 0 (0)
Bilirubin associated with graft versus host disease (GVHD) (Investigations) | 5 (5) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC (Investigations) | 3 (3) | 0 (0)
Infection, Bacterial (Infections and infestations) | 13 (13) | 0 (0)
Infection, Fungal (Infections and infestations) | 3 (3) | 0 (0)
Infection, Viral (Infections and infestations) | 8 (8) | 0 (0)
Lymphatics (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 31 (31) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 23 (23) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 25 (25) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 11 (11) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 8 (8) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 20 (20) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 23 (23) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 20 (20) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 24 (24) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 27 (27) | 0 (0)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 21 (21) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 16 (16) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 15 (15) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration (Nervous system disorders) | 11 (11) | 0 (0)
Neurology - Other (Nervous system disorders) | 4 (4) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 3 (3) | 0 (0)
Speech impairment (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 12 (12) | 0 (0)
Dry eye syndrome (Eye disorders) | 2 (2) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 4 (4) | 0 (0)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 25 (25) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes